CLINICAL TRIAL: NCT06820736
Title: A Prospective, Randomized Comparison Of Drainage Techniques After One- Or Two-Level Open Posterior Lumbar Decompression Or Decompression And Fusion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Twin Cities Spine Center (Other)
Collaborators: Allina Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2199368-6
Record Dates: First submitted 2025-02-05; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Complications, Postoperative
Keywords: Lumbar spine surgery; drain; postoperative complications
MeSH Terms: conditions — Postoperative Complications | interventions — Drainage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Active Drain (Experimental): The drain will be used with compression suction.
  Interventions: Device: Drain
- Passive Drain (Experimental): The drain will be used with gravity alone.
  Interventions: Device: Drain
- No Drain (No Intervention): No drain will be used.

INTERVENTIONS:
Device: Drain — A drain is a small flexible tube that is placed next to where the spine was operated upon.
  Arms: Active Drain; Passive Drain

SUMMARY:
This project is being done to understand if a drain reduces recovery problems after surgery, such as infection or the need for more surgery.

DETAILED DESCRIPTION:
The primary objective is to prospectively evaluate drains used in lumbar spine surgery in patients undergoing one- or two-level open posterior lumbar decompression or decompression and fusion for the relative risk of return to the operating room within 90 days.

ELIGIBILITY:
Inclusion Criteria:

* One or two-level open spinal decompression or decompression and fusion for the treatment of lumbar stenosis and/or spondylolisthesis

Exclusion Criteria:

* Infection, tumor, or trauma
* Prior lumbar fusion surgery
* Lumbar fusion surgery at more than 2 levels
* Anterior lumbar surgery
* Perioperative anticoagulation treatment
* Intraoperative incidental durotomy
* Intraoperative or postoperative cerebrospinal fluid leakage
* Intraoperative EBL greater than one liter

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 975 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2035-01-09 (Estimated); Study Completion 2040-01-09 (Estimated)

PRIMARY OUTCOMES:
Reoperation | 90 days postoperatively
  Relative risk of return to the operating room

SECONDARY OUTCOMES:
Time to drain removal | 90 days postoperatively
  Time (minutes) to drain removal
Drain volume | 90 days postoperatively
  Daily volume (mL) of fluid collected by the drain
Transfusion | 90 days postoperatively
  Need (yes or no) for a postoperative transfusion
Length of Stay | 90 days postoperatively
  Length of hospital stay
Complications | 90 days postoperatively
  Occurrence (yes/no) of wound complications, wound dehiscence, superficial wound infection or deep wound inflection

CONTACTS AND LOCATIONS:
Overall Officials: Ben Mueller, MD, PhD, Principal Investigator — Twin Cities Spine Center
Locations (1):
- Abbott Northwestern Hospital, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
We do not want to share IPD

REFERENCES:
- [Background] Reier L, Fowler JB, Arshad M, Siddiqi J. Drains in Spine Surgery for Degenerative Disc Diseases: A Literature Review to Determine Its Usage. Cureus. 2022 Mar 13;14(3):e23129. doi: 10.7759/cureus.23129. eCollection 2022 Mar. PMID 35464540
- [Background] Davidoff CL, Rogers JM, Simons M, Davidson AS. A systematic review and meta-analysis of wound drains in non-instrumented lumbar decompression surgery. J Clin Neurosci. 2018 Jul;53:55-61. doi: 10.1016/j.jocn.2018.04.038. Epub 2018 Apr 19. PMID 29680443
- [Background] Patel SB, Griffiths-Jones W, Jones CS, Samartzis D, Clarke AJ, Khan S, Stokes OM. The current state of the evidence for the use of drains in spinal surgery: systematic review. Eur Spine J. 2017 Nov;26(11):2729-2738. doi: 10.1007/s00586-017-4983-0. Epub 2017 Feb 11. PMID 28190206
- [Background] Zijlmans JL, Buis DR, Verbaan D, Vandertop WP. Wound drains in non-complex lumbar surgery: a systematic review. Bone Joint J. 2016 Jul;98-B(7):984-9. doi: 10.1302/0301-620X.98B7.37190. PMID 27365478
- [Background] Liu Y, Li Y, Miao J. Wound drains in posterior spinal surgery: a meta-analysis. J Orthop Surg Res. 2016 Jan 22;11:16. doi: 10.1186/s13018-016-0351-8. PMID 26801088
- [Background] Liu JM, Chen WZ, Fu BQ, Chen JW, Liu ZL, Huang SH. The Use of Closed Suction Drainage in Lumbar Spinal Surgery: Is It Really Necessary? World Neurosurg. 2016 Jun;90:109-115. doi: 10.1016/j.wneu.2016.02.091. Epub 2016 Mar 2. PMID 26944885
- [Background] Mirzai H, Eminoglu M, Orguc S. Are drains useful for lumbar disc surgery? A prospective, randomized clinical study. J Spinal Disord Tech. 2006 May;19(3):171-7. doi: 10.1097/01.bsd.0000190560.20872.a7. PMID 16770213
- [Background] Walid MS, Abbara M, Tolaymat A, Davis JR, Waits KD, Robinson JS 3rd, Robinson JS Jr. The role of drains in lumbar spine fusion. World Neurosurg. 2012 Mar-Apr;77(3-4):564-8. doi: 10.1016/j.wneu.2011.05.058. Epub 2011 Nov 7. PMID 22120372
- [Background] Kanayama M, Oha F, Togawa D, Shigenobu K, Hashimoto T. Is closed-suction drainage necessary for single-level lumbar decompression?: review of 560 cases. Clin Orthop Relat Res. 2010 Oct;468(10):2690-4. doi: 10.1007/s11999-010-1235-6. Epub 2010 Jan 21. PMID 20091386
- [Background] Scuderi GJ, Brusovanik GV, Fitzhenry LN, Vaccaro AR. Is wound drainage necessary after lumbar spinal fusion surgery? Med Sci Monit. 2005 Feb;11(2):CR64-6. PMID 15668633
- [Background] Brown MD, Brookfield KF. A randomized study of closed wound suction drainage for extensive lumbar spine surgery. Spine (Phila Pa 1976). 2004 May 15;29(10):1066-8. doi: 10.1097/00007632-200405150-00003. PMID 15131430
- [Background] Payne DH, Fischgrund JS, Herkowitz HN, Barry RL, Kurz LT, Montgomery DM. Efficacy of closed wound suction drainage after single-level lumbar laminectomy. J Spinal Disord. 1996 Oct;9(5):401-3. PMID 8938608
- [Background] Smith VA, Coffman CJ, Hudgens MG. Interpreting the Results of Intention-to-Treat, Per-Protocol, and As-Treated Analyses of Clinical Trials. JAMA. 2021 Aug 3;326(5):433-434. doi: 10.1001/jama.2021.2825. No abstract available. PMID 34342631
- [Background] Pourhoseingholi MA, Vahedi M, Rahimzadeh M. Sample size calculation in medical studies. Gastroenterol Hepatol Bed Bench. 2013 Winter;6(1):14-7. PMID 24834239
- [Background] Porto GBF, Jeffrey Wessell DO, Alvarado A, Arnold PM, Buchholz AL. Anticoagulation and Spine Surgery. Global Spine J. 2020 Jan;10(1 Suppl):53S-64S. doi: 10.1177/2192568219852051. Epub 2020 Jan 6. PMID 31934522
- [Background] Horlocker TT, Nuttall GA, Dekutoski MB, Bryant SC. The accuracy of coagulation tests during spinal fusion and instrumentation. Anesth Analg. 2001 Jul;93(1):33-8. doi: 10.1097/00000539-200107000-00008. PMID 11429335
- [Background] Tomasino A, Lumenta CB. To drain or not to drain: about using wound drainage after instrumented spine procedures. World Neurosurg. 2012 Mar-Apr;77(3-4):466-7. doi: 10.1016/j.wneu.2011.07.035. Epub 2011 Nov 7. No abstract available. PMID 22120318
- [Background] Butler AJ, Donnally CJ 3rd, Goz V, Basques BA, Vaccaro AR, Schroeder GD. Symptomatic Postoperative Epidural Hematoma in the Lumbar Spine. Clin Spine Surg. 2022 Nov 1;35(9):354-362. doi: 10.1097/BSD.0000000000001278. Epub 2021 Dec 20. PMID 34923504
- [Background] Chen Q, Zhong X, Liu W, Wong C, He Q, Chen Y. Incidence of postoperative symptomatic spinal epidural hematoma requiring surgical evacuation: a systematic review and meta-analysis. Eur Spine J. 2022 Dec;31(12):3274-3285. doi: 10.1007/s00586-022-07421-6. Epub 2022 Oct 19. PMID 36260132
- [Background] Sokolowski MJ, Garvey TA, Perl J 2nd, Sokolowski MS, Cho W, Mehbod AA, Dykes DC, Transfeldt EE. Prospective study of postoperative lumbar epidural hematoma: incidence and risk factors. Spine (Phila Pa 1976). 2008 Jan 1;33(1):108-13. doi: 10.1097/BRS.0b013e31815e39af. PMID 18165756